CLINICAL TRIAL: NCT04027192
Title: Randomized, Placebo-controlled, Double-blind, Parallel Group Study to Investigate Safety, Tolerability and Pharmacokinetics of Increasing Multiple Oral Doses of BAY2328065 Including the CYP3A4 Induction Potential of BAY2328065 and Randomized Cross-over Investigation of the Relative Bioavailability Between Solution and Tablet Formulation in Healthy Male Participants
Brief Title: Study to Test the Safety of Increasing Multiple Doses of BAY2328065 Given by Mouth, How the Drug is Tolerated and Acts in the Human Body of Healthy Male Participants. Alteration of the Study Drug Effects by Another Drug and the Availability of the Drug Given in Different Formulations is Also Tested.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 19251; 2019-000940-90 (EudraCT Number)
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: The study will be performed in 2 study parts. Each participant will take part in one study part only.
  * Bridging part: This will be a single-center, randomized, open-label cross-over part with 3 study interventions, 3 intervention periods and 2 intervention sequences.
  * Multiple dose escalation part: This will be a single-center, randomized, placebo-controlled, double-blind, parallel group multiple dose escalation part.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open-label crossover in bridging part; double-blind, parallel group in multiple dose escalation part
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Bridging part: intervention sequence ABC or BAC (Experimental): 10 healthy male participants will be randomly allocated to this arm. The study interventions will follow the sequence ABC or BAC: A: single dose of 50 mg BAY2328065 given as LSF in fasted state B: single dose of 50 mg BAY2328065 given as tablet in fasted state C: single dose of 50 mg BAY2328065 given as tablet in fed state (i.e. after a high caloric and high fat meal)
  Interventions: Drug: BAY2328065 LSF; Drug: BAY2328065 tablet
- Multiple dose escalation part: dose 1 (Experimental): 10 participants will be randomly allocated to active drug or placebo (8 active drug, 2 placebo).
  The study intervention will be administered with a single dose on the first dosing day followed by twice daily doses for 10 days followed by a single dose on the last dosing day
  Interventions: Drug: BAY2328065 LSF; Drug: Placebo LSF
- Multiple dose escalation part: dose 2 (Experimental): 10 participants will be randomly allocated to active drug or placebo (8 active drug, 2 placebo).
  The study intervention will be administered with a single dose on the first dosing day followed by twice daily doses for 10 days followed by a single dose on the last dosing day Midazolam is given for investigation of drug-drug interaction
  Interventions: Drug: BAY2328065 tablet; Drug: Placebo tablet; Drug: Midazolam
- Multiple dose escalation part: dose 3 (Experimental): 10 participants will be randomly allocated to active drug or placebo (8 active drug, 2 placebo).
  The study intervention will be administered with a single dose on the first dosing day followed by twice daily doses for 10 days followed by a single dose on the last dosing day Midazolam is given for investigation of drug-drug interaction
  Interventions: Drug: BAY2328065 tablet; Drug: Placebo tablet; Drug: Midazolam
- Multiple dose escalation part: dose 4 (Experimental): 10 participants will be randomly allocated to active drug or placebo (8 active drug, 2 placebo).
  The study intervention will be administered with a single dose on the first dosing day followed by twice daily doses for 10 days followed by a single dose on the last dosing day Midazolam is given for investigation of drug-drug interaction
  Interventions: Drug: BAY2328065 tablet; Drug: Placebo tablet; Drug: Midazolam
- Multiple dose escalation part: dose 5 (Experimental): 10 participants will be randomly allocated to active drug or placebo (8 active drug, 2 placebo).
  The study intervention will be administered with a single dose on the first dosing day followed by a treatment pause of 2 days followed by twice daily doses for 1 day followed by three times daily doses for 9 days followed by a single dose on the last dosing day Midazolam is given for investigation of drug-drug interaction
  Interventions: Drug: BAY2328065 tablet; Drug: Placebo tablet; Drug: Midazolam

INTERVENTIONS:
Drug: BAY2328065 LSF — 20 mg/mL LSF (liquid service formulation), orally
  Arms: Bridging part: intervention sequence ABC or BAC; Multiple dose escalation part: dose 1
Drug: BAY2328065 tablet — 50 mg tablet, orally
  Arms: Bridging part: intervention sequence ABC or BAC; Multiple dose escalation part: dose 2; Multiple dose escalation part: dose 3; Multiple dose escalation part: dose 4; Multiple dose escalation part: dose 5
Drug: Placebo LSF — Matching Placebo LSF, orally
  Arms: Multiple dose escalation part: dose 1
Drug: Placebo tablet — Matching Placebo tablet, orally
  Arms: Multiple dose escalation part: dose 2; Multiple dose escalation part: dose 3; Multiple dose escalation part: dose 4; Multiple dose escalation part: dose 5
Drug: Midazolam — 1 mg per day, orally
  Arms: Multiple dose escalation part: dose 2; Multiple dose escalation part: dose 3; Multiple dose escalation part: dose 4; Multiple dose escalation part: dose 5

SUMMARY:
Study on the safety and tolerability of a new drug BAY2328065 when given increased doses as tablet or solution over 12 days to healthy male participants. Researcher want to study how the body absorbs, breaks down and excrete the new drug, also when given together with a test meal. In addition the study will investigate changes that take place in the body when BAY2328065 is given together with another drug.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, ECG and vital signs
* Confirmation of the subject's health insurance coverage prior to the first screening examination/visit
* Body mass index (BMI) within the range 18 and 30 kg/m^2 (inclusive)
* Male participants who are sexually active must agree to use two reliable and acceptable methods of contraception simultaneously (one method used by the study participant and one method used by the partner) and not to act as sperm donor until follow-up
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* The informed consent must be signed before any study specific tests or procedures are done
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention will not be normal
* Relevant diseases within the last 4 weeks prior to start of the first study intervention
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Existing chronic diseases requiring medication
* History of cardiovascular disease
* Known diseases as specified in protocol
* Regular use of therapeutic or recreational drugs
* Suspicion of drug or alcohol abuse
* Smoking equal or more than 10 cigarettes/day
* Clinically relevant findings in Electrocardiogram (ECG), blood pressure, heart rate, physical examination, laboratory examination
* History of COVID-19
* Contact with SARS-CoV-2 positive persons or COVID-19 patients within the last 4 weeks prior admission to the ward
* Positive SARS-CoV-2 viral RNA test

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) | From first dosing up to 30 days after end of treatment with study intervention, summing up to approximately 39 to 45 days for a participant
Severity of TEAEs | From first dosing up to 30 days after end of treatment with study intervention, summing up to approximately 39 to 45 days for a participant
AUC(0-12)md (twice daily [BID]) | From first dose of BAY2328065 until 72 hour after the last dose of BAY2328065
Cmax,md of BAY2328065 | From first dose of BAY2328065 until 72 hour after the last dose of BAY2328065

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.